CLINICAL TRIAL: NCT00188734
Title: Lung Cancer Screening in High-risk Smokers Using Low-dose Computed Tomography
Brief Title: Early Lung Cancer Detection Using Computed Tomography
Status: Completed | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: I-ELCAP
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Last update posted 2016-08-10 (Estimated); Status verified 2016-08

CONDITIONS: Lung Cancer
Keywords: Lung Cancer; Eary Diagnosis; Screening
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
Early detection of lung cancer may improve treatment outcomes. Risk factors have been identified, suggesting a population which might benefit from regular screening. Lung cancer screening using low-dose computed tomography (LDCT) has experienced a recent renaissance with reported sensitivity for detection of lung cancer of 2.7% in high-risk populations. The purpose of this study is to evaluate the utility of LCDT for the early diagnosis of lung cancer in Ontario.

ELIGIBILITY:
Inclusion Criteria:

55 years or older at least 10 pack-year history of smoking general good health

Exclusion Criteria:

any prior cancers except non-melanotic skin cancer

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: high risk current and former smokers
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Actual)
Dates: Start 2003-09; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Heidi C Roberts, MD, Principal Investigator — University Health Network, Toronto
Locations (1):
- Princess Margaret Hospital, Toronto, Ontario, Canada